CLINICAL TRIAL: NCT05579717
Title: Examining the Effectiveness of Equine Assisted Learning for Trauma-exposed Public Safety Personnel
Brief Title: Examining the Effectiveness of EAL
Acronym: EAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: University of Saskatchewan (Other); University of Regina (Other)
Responsible Party: Principal Investigator, Margaret McKinnon, Professor, McMaster University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14547
Record Dates: First submitted 2022-09-28; First posted 2022-10-14 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Trauma
Keywords: EAL; PTSD; posttraumatic stress disorder; public safety personnel; first responder; Equine Assisted Learning; horse therapy; trauma
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to an intervention group or a waitlist control group based on the time they complete their initial baseline interview. Individuals in the waitlist control group will be offered the opportunity to participate in EAL once they have completed the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Equine Assisted Learning group (Experimental): Participants in this group will receive 16 sessions of Equine Assisted Learning (EAL), facilitated by a trained clinician at Cartier Farms.
  Interventions: Behavioral: Equine Assisted Learning
- Waitlist control group (No Intervention): Participants in the waitlist control group will not receive EAL for the duration of the study.

INTERVENTIONS:
Behavioral: Equine Assisted Learning — EAL is an intervention in which mental health clinicians and equine specialists work together with clients to address a learning goal via unmounted interaction with a horse. It is 16 sessions in length, at a rate of two sessions per week.
  Other Names: EAL
  Arms: Equine Assisted Learning group

SUMMARY:
This quasi-experiment will evaluate the effectiveness of Equine Assisted Learning for reducing symptoms associated with trauma exposure among public safety personnel (e.g., fire fighters, police, paramedics, etc.).

DETAILED DESCRIPTION:
The purpose of the proposed project is to investigate the effectiveness of Equine Assisted Learning (EAL) for reducing symptoms associated with trauma exposure among public safety personnel. EAL is an intervention in which mental health clinicians and equine specialists work together with clients to address a learning goal via unmounted interaction with a horse. Recent literature indicates that EAL shows promise in addressing a range of mental health diagnoses among a variety of populations, including military and Royal Canadian Mounted Police veterans with PTSD. The EAL intervention will be delivered at Cartier Farms in Spruce Home, Saskatchewan. Research components of this study will be conducted virtually via Zoom.

The investigators will employ a quasi-experimental design with pre-post and follow-up testing. Participants will be assigned one of two groups based on the time that they complete their initial baseline interview: (1) the intervention group will receive the EAL intervention for 8 weeks, while (2) the waitlist control condition will not receive this treatment for the same amount of time. Data on trauma exposure symptom severity will be collected from all participants prior to the start of the the study (baseline), again 8 weeks later (post), and then a final time 3 months later (follow-up). The two conditions will then be compared to determine whether there are differences in trauma exposure symptom severity between groups. To obtain a sufficient sample size while also running appropriately sized interventions of 6-10 participants per session, the researchers will conduct 4-6 rounds of group assignment. All individuals in the waitlist control condition will be offered EAL following their completion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking adults;
2. Currently or previously employed as public safety personnel (e.g., police officer, fire fighter, paramedic, healthcare worker, emergency dispatcher, correctional officer);
3. Reside in Saskatchewan;
4. Meet diagnostic criteria for having experienced a Criterion A traumatic event;
5. Able to provide written informed consent;
6. Have access to a smart phone, tablet, or computer with a working microphone and camera; and
7. Have access to consistent and reliable internet.

Exclusion:

1. Meet/met current/past diagnostic criteria for several psychiatric, neurodevelopmental, and neurological conditions;
2. History of severe head trauma with loss of consciousness or history of traumatic brain injury;
3. Have previously completed at least half of the EAL curriculum at Cartier Farms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
PTSD symptomatology | 20 weeks
  Changes in performance on the Clinician Administered PTSD Scale (structured interview) at pre, post, and follow-up.
PTSD symptomatology | 20 weeks
  Changes in performance on the PTSD Checklist for DSM-5 at pre, post, and follow-up. Scores can range between 0 and 80 with higher scores denoting higher PTSD symptomatology.

SECONDARY OUTCOMES:
Mental health symptomatology | 20 weeks
  Changes in performance on the Mini International Neuropsychiatric Interview (structured interview) at pre, post, and follow-up.
Depression, anxiety, and stress symptomatology | 20 weeks
  Changes in performance on the Depression Anxiety Stress Scale at pre, post, and follow-up. Scores can range between 0 and 42 with higher scores denoting higher depression, anxiety, and/or stress symptomatology.
Substance involvement | 20 weeks
  Changes in performance on the World Health Organization's Alcohol, Smoking, and Substance Involvement Test at pre, post, and follow-up. Each question on the ASSIST has a checklist set of responses to choose from to measure substances used in the past, and each response from questions 2 to 7 has a numerical score. Higher scores indicate more significant substance involvement.
Health complaints | 20 weeks
  Changes in performance on the Physical Symptoms Questionnaire at pre, post, and follow-up. Scores can range between 0 and 33 with higher scores denoting more health complaints.
Sleep quality | 20 weeks
  Changes in performance on the Pittsburgh Sleep Quality Index at pre, post, and follow-up. Scores can range between 0 and 21 with higher scores denoting poorer sleep quality.
Body awareness | 20 weeks
  Changes in performance on the Multidimensional Assessment of Interoceptive Awareness - Version 2 at pre, post, and follow-up. Scores can range between 0 and 185 with higher scores denoting greater body awareness.
Moral injury | 20 weeks
  Changes in performance on the Moral Injury Assessment - Public Safety Personnel at pre, post, and follow-up. Scores can range between 17 and 102 with higher scores denoting higher moral injury.
Dissociation | 20 weeks
  Changes in performance on the Multiscale Dissociation Index at pre, post, and follow-up. Scores can range between 0 and 120 with higher scores denoting higher dissociative symptomatology.
Emotion regulation | 20 weeks
  Changes in performance on the Difficulties in Emotion Regulation Scale, at pre, post, and follow-up. Scores can range between 36 and 180 with higher scores denoting poorer emotion regulation.
Exposure to childhood trauma | Completed once at baseline
  Baseline description of trauma experienced in childhood based on the Childhood Trauma Questionnaire, which is a 28-item checklist where more endorsed traumatic experiences indicates more exposure to childhood trauma.
Alcohol use disorder symptomatology | 20 weeks
  Changes in performance on the Alcohol Use Disorder Identification Test at pre, post, and follow-up. Scores can range between 0 and 40 with higher scores denoting higher AUD symptomatology.
Cannabis use disorder symptomatology | 20 weeks
  Changes in performance on the Cannabis Use Disorder Identification Test at pre, post, and follow-up. Scores can range between 0 and 32 with higher scores denoting higher CUD symptomatology.
Substance use disorder symptomatology | 20 weeks
  Changes in performance on the Drug Use Disorder Identification Test at pre, post, and follow-up. Scores can range between 0 and 44 with higher scores denoting higher SUD symptomatology.
Resilience | 20 weeks
  Changes in performance on the Brief Resilience Scale at pre, post, and follow-up. Scores can range between 6 and 30 with higher scores denoting higher resilience.
Self-compassion | 20 weeks
  Changes in performance on the Self Compassion Scale at pre, post, and follow-up. Scores can range between 26 and 130 with higher scores denoting higher self-compassion.
Health and disability | 20 weeks
  Changes in performance on World Health Organization's Disability Assessment Schedule 12 at pre, post, and follow-up. Scores can range between 0 and 100 with higher scores denoting greater disability.
Disability | 20 weeks
  Changes in performance on the Sheehan Disability Scale at pre, post, and follow-up. Scores can range between 0 and 44 with higher scores denoting greater disability.
Work functioning and productivity | 20 weeks
  Changes in performance on Lam's Employment and Productivity Scale at pre, post, and follow-up. Scores can range between 0 and 28 with higher scores denoting more severe work impairment.

OTHER OUTCOMES:
Heart rate variability | 20 weeks
  Changes in heart rate variability over time, as measured by a Garmin VivoActive 4 smartwatch.
Sleep quality | 20 weeks
  Changes in sleep quality over time, as measured by a Garmin VivoActive 4 smartwatch.
Experience in EAL | 8 weeks
  Participant experience in EAL as measured by a semi-structured, qualitative interview.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret McKinnon, PhD, CPsych, Principal Investigator — McMaster University
Locations (1):
- Cartier Farms, Prince Albert, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No